CLINICAL TRIAL: NCT06060236
Title: Comparison of Analgesic Efficacy of Dexketoprofen and Ibuprofen in Long Bone Fractures: Randomised Controlled Double-blind Study
Brief Title: Dexketoprofen and Ibuprofen in Long Bone Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Safa Dönmez, Department of Emergency Medicine, M.D. Specialist, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2-23-4743
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Pain; Bone Fracture
Keywords: Long bone fracture; ibuprofen; dexketoprofen; pain
MeSH Terms: conditions — Pain; Fractures, Bone | interventions — Ibuprofen; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ibuprofen (Experimental): ibuprofen intravenous 800 mg
  Interventions: Drug: Ibuprofen 800 mg
- dexketoprofen (Experimental): dexketoprofen intravenous 50 mg
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Ibuprofen 800 mg — Ibuprofen 800 Mg İv
  Arms: ibuprofen
Drug: Dexketoprofen — Dexketoprofen 50 Mg İV
  Arms: dexketoprofen

SUMMARY:
The aim of this study was to compare the efficacy of ibuprofen and dexketoprofen, two common analgesic drugs used in pain control in patients with long bone fractures.

DETAILED DESCRIPTION:
Long bone fractures are the fractures of long bones (tibia, femur, humerus) in the human body. Such fractures usually occur as a result of trauma and are manifested by symptoms such as pain, swelling, bruising and limitation of movement. Effective control of pain can help the patient relax and facilitate the healing process. Ibuprofen and dexketoprofen, which belong to the class of non-steroidal anti-inflammatory drugs (NSAID), are among the analgesics commonly used in the pain management of all fractures. These drugs are thought to be able to relieve pain, reduce inflammation, and help patients move. However, each patient's individual response and tolerance may differ, so the efficacy and side effects of each drug may vary from patient to patient. This makes it difficult to determine which analgesic is more effective and safe in clinical practice. The fact that it is a subject that has not been done much in the literature has led us to do this study.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* Patients under 80 years of age
* Patients who agreed to participate in the study
* One of the tibia, femur and humerus bones is broken
* Patients with a VAS score of 50 and above
* Patients with no other injuries requiring emergency surgery
* Previously known adverse reactions to the active ingredient of the drugs to be used patients with no history
* Conscious patients
* Oriented cooperative patients

Exclusion Criteria:

* Patients under the age of 18 and over the age of 80
* Patients who did not agree to participate in the study
* Patients with vital signs outside the normal limits
* Patients with a history of adverse reactions to known NSAIDs
* Those who cannot determine the severity of pain on the VAS
* Patients with a VAS Score of 50 mm or less
* Those with other orthopedic injuries pregnant women
* Those with advanced systemic disease
* Those with malignancy
* Those with chronic liver and kidney disease
* Those who use neuro-psychiatric drugs with sedative and analgesic effects
* Those with a history of psychological and neurological diseases
* Patients using analgesics 8 hours before the examination

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | 120 minute
  The pain is determined using a 100 mm scale. Patients are instructed to mark the level of pain they experience, with 0 mm indicating no pain and 100 mm indicating the presence of maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Safa Dönmez, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent Şehir Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Poonai N, Bhullar G, Lin K, Papini A, Mainprize D, Howard J, Teefy J, Bale M, Langford C, Lim R, Stitt L, Rieder MJ, Ali S. Oral administration of morphine versus ibuprofen to manage postfracture pain in children: a randomized trial. CMAJ. 2014 Dec 9;186(18):1358-63. doi: 10.1503/cmaj.140907. Epub 2014 Oct 27. PMID 25349008
- [Result] Friday JH, Kanegaye JT, McCaslin I, Zheng A, Harley JR. Ibuprofen provides analgesia equivalent to acetaminophen-codeine in the treatment of acute pain in children with extremity injuries: a randomized clinical trial. Acad Emerg Med. 2009 Aug;16(8):711-6. doi: 10.1111/j.1553-2712.2009.00471.x. Epub 2009 Jul 14. PMID 19624576